CLINICAL TRIAL: NCT04053426
Title: Agitation Follow up After Introduction of a New Patient Care Algorithm
Acronym: SARA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.344; 2018-A00582-53 (Other: ID RCB)
Record Dates: First submitted 2019-07-01; First posted 2019-08-12 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Agitation,Psychomotor
Keywords: RASS; CAM-ICU
MeSH Terms: conditions — Psychomotor Agitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population "before": Patient included before implementation of care algorithm.
- Population "after": Patients included after the implementation of care algorithm and training of health professionnals
  Interventions: Other: Implementation of agitation care algorithm

INTERVENTIONS:
Other: Implementation of agitation care algorithm — Following the agitation care algorithm care professional adapt their behavior regarding agitation
  Groups: Population "after"

SUMMARY:
Agitation in the intensive care unit is motor hyperactivity. It is frequent (b/w 30% to 70%) and has multiple causes: pain, medical reason, delirium, medication, etc. It can be a source of complication, for the patient, and equipment pullout. International recommendations state that the agitation should be taken care of with standardized protocols to improve patient care.

DETAILED DESCRIPTION:
Data regarding patient characteristics and evaluation criterion will be collected automatically with the unit software (CCC, General Electrics) in specific file.

Care and health teams enter the data systematically following the usual protocol.

First Step :

Follow-up and collection of data of patients included. Agitation evaluation with RASS scale, pain evaluation with BPS or NPRS.

Second Step:

Team training to delirium evaluation scale (CAM-ICU) and to the use of care algorithm.

Third Step:

Follow-up and collection of data of patients included. Use of care algorithm by doctors, nurses and back up training nurse to ensure daily information to health professionals of the care unit.

Concomitant Step:

Post discharge from care unit medical appointment to evaluate anxiety symptoms (HAD scale) and quality of life (SF-12)

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting an agitation episode (RASS>1)
* Intensive care unit hospitalization
* Patient or next of kin if patient not able non opposed on participating to the study

Exclusion Criteria:

* Decision to limit life-sustaining therapy
* Brain damage
* Moribund patient
* Patient participating to another trial excluding observational studies
* The patient is pregnant or a lactating female
* Patient under tutorship or curatorship and liberty deprived

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in the intensive care unit requiring and presenting a first episode of agitation.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
RASS scale evaluation between phase "before" and phase "after" | at the end of each phase, average of 1 year
  Comparison of the duration of agitation between phase "before" and phase "after"

CONTACTS AND LOCATIONS:
Overall Officials: Claire Chapuis, Dr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chanques G, Jaber S, Barbotte E, Violet S, Sebbane M, Perrigault PF, Mann C, Lefrant JY, Eledjam JJ. Impact of systematic evaluation of pain and agitation in an intensive care unit. Crit Care Med. 2006 Jun;34(6):1691-9. doi: 10.1097/01.CCM.0000218416.62457.56. PMID 16625136
- [Background] Almeida TM, Azevedo LC, Nose PM, Freitas FG, Machado FR. Risk factors for agitation in critically ill patients. Rev Bras Ter Intensiva. 2016 Oct-Dec;28(4):413-419. doi: 10.5935/0103-507X.20160074. PMID 28099638
- [Background] Jaber S, Chanques G, Altairac C, Sebbane M, Vergne C, Perrigault PF, Eledjam JJ. A prospective study of agitation in a medical-surgical ICU: incidence, risk factors, and outcomes. Chest. 2005 Oct;128(4):2749-57. doi: 10.1378/chest.128.4.2749. PMID 16236951
- [Background] Reade MC, Finfer S. Sedation and delirium in the intensive care unit. N Engl J Med. 2014 Jan 30;370(5):444-54. doi: 10.1056/NEJMra1208705. No abstract available. PMID 24476433
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Payen JF, Bosson JL, Chanques G, Mantz J, Labarere J; DOLOREA Investigators. Pain assessment is associated with decreased duration of mechanical ventilation in the intensive care unit: a post Hoc analysis of the DOLOREA study. Anesthesiology. 2009 Dec;111(6):1308-16. doi: 10.1097/ALN.0b013e3181c0d4f0. PMID 19934877
- [Background] Payen JF, Chanques G, Mantz J, Hercule C, Auriant I, Leguillou JL, Binhas M, Genty C, Rolland C, Bosson JL. Current practices in sedation and analgesia for mechanically ventilated critically ill patients: a prospective multicenter patient-based study. Anesthesiology. 2007 Apr;106(4):687-95; quiz 891-2. doi: 10.1097/01.anes.0000264747.09017.da. PMID 17413906
- [Background] Ely EW, Stephens RK, Jackson JC, Thomason JW, Truman B, Gordon S, Dittus RS, Bernard GR. Current opinions regarding the importance, diagnosis, and management of delirium in the intensive care unit: a survey of 912 healthcare professionals. Crit Care Med. 2004 Jan;32(1):106-12. doi: 10.1097/01.CCM.0000098033.94737.84. PMID 14707567